CLINICAL TRIAL: NCT05072496
Title: A Prospective Cohort Study on Antibody Persistence and Immune Memory After Two Doses of Inactivated COVID-19 Vaccine in 150 People
Brief Title: Study on Antibody Persistence and Immune Memory of Inactivated COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Wu Jiang, Director of Institute for Vaccines and Immunization, Centers for Disease Control and Prevention, China
Other Study IDs: BJCDCWJ202101
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: Inactivated vaccine; cohort study; Antibody persistence; cellular immunity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study describe 1 year durability of humoral and cellular immune responses in 150 individuals who received COVID-19 inactivated vaccine. all participants were recruited aged between 18 and 59 years old. Every participant was familiarized with the aim of the study and asked to sign an informed consent agreement, and be required blood sampling at the day 0 of first dose vaccine and 1 month, 3 months, 6 months and 12 months after fully vaccination separately. From every sample, 10 ml, 10 ml, and 5 ml were dispensed in three vacuum blood collection tubes. Peripheral blood lymphocytes cell (PBMC) were isolated with the two 10 ml samples contained heparin to detect immune memory cells and cytokines. RBD-IgG and neutralizing antibody be detected by 5ml sample from separating gel vacuum tubes. every individual conducted a detailed analysis comparing neutralizing antibody, TEM, TCM , and report on the cellular and humoral immunity 1 year after accept COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Working at the CDC
* Between the ages of 18 and 59
* Healthy
* Not vaccinated with COVID-19 vaccine
* Agreed to take a blood sample

Exclusion Criteria:

* who cannot take the COVID-19 vaccine due to some personal reasons
* history of SARS-CoV, SARS-CoV-2, or Middle East respiratory syndrome infection
* high-risk epidemiology history within 14 days before enrolment (eg, travel or residence history in communities with case reports, or contact history with someone infected with SARS-CoV-2)
* axillary temperature of more than 37·0℃
* history of allergy to any vaccine component.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The healthy people aged between 18 and 59, and have not been infected with COVID-19, have not been vaccinated with COVID-19 vaccine, and agree to collect blood samples.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Durability of humoral and cellular immune responses | 12 months after fully vaccination
  The humoral immunogenicity outcomes include the RBD-specific IgG titers and neutralising antibodies amounts at 1, 3, 6, and 12 months after the second shot. The positive cutoff for RBD-specific IgG antibodies was defined as the sample cutoff (S/CO) value ≥1.0. Seroconversion of neutralising antibodies was defined as a change from seronegative at baseline to seropositive or a four-fold titre increase. The positive cutoff of the titre for neutralising antibodies was 1/4.
  The cellular immune response outcomes measured by ICS assays across the blood collection time points.the percentage of RBD-specific CD4+ CD8+ memory T cells after vaccination.

SECONDARY OUTCOMES:
The dynamic variation of the level of antibody | 1，3，6 , 12 month
  RBD-IgG and neutralizing antibody level after vaccination at 1,3 and 6 ,12months vaccination.
Cytokine secretion by peripheral blood mononuclear cells | 1,3,6,12 month
  To study the cytokine production of PBMC after stimulation with RBD after vaccination at 1,3,6 and 12 months vaccination,for examples IL-2,IL-5,IFN and GrB.
TCM and TEM amount varies at different time points | 1,3,6,12 month
  The dynamic variation of specificity TCM and TEM after vaccination at 1,3,6 and 12 months vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Center for Disease Control and Prevention, Beijing, China